CLINICAL TRIAL: NCT02617797
Title: Radiofrequency in the Female Stress Urinary Incontinence: A Randomized Clinical Trial
Brief Title: Radiofrequency in the Female Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1162-0945
Record Dates: First submitted 2015-11-22; First posted 2015-12-01 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Urinary Stress Incontinence
Keywords: Urinary Stress Incontinence; Radiofrequency; Women
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency (Experimental): Experimental group: women with urinary incontinence are subjected to standard treatment kinesiotherapy perineal ( pelvic muscle exercises ) every day in home and one session per week in the clinic in beyond the RF application in the genital area once a week to total 5 sessions.
  Interventions: Device: Radiofrequency
- Radiofrequency Off (Sham Comparator): Control group: women with stress urinary incontinence will be submitted to the treatment of kinesiotherapy standard perineal ( pelvic muscle exercises ) every day in home and one session per week in the clinic beyond the application of radiofrequency off in genital area once a week with the total of 5 sessions.
  Interventions: Device: Radiofrequency OFF

INTERVENTIONS:
Device: Radiofrequency — The radiofrequency is a noninvasive technique that will be applied to the external urethral meatus region.It will use a digital thermometer with infrared to mention the temperature should reach 39 ° C and maintain this temperature for 2 minutes.It will use a digital thermometer with infrared to mention the temperature should reach 39 ° C and maintain this temperature for 2 minutes
  Arms: Radiofrequency
Device: Radiofrequency OFF — Will be used to put off radio frequency will be heated glycerin to occur masking for the patient.
  Arms: Radiofrequency Off

SUMMARY:
Urinary stress incontinence ( SUI ) is defined as an involuntary loss of urinary Complaint no effort According to the Consensus of the International Continence Society (Society Continence International - ICS) . SUI Prevalence of adult female Population and 25 % to 30 %.However, despite the high prevalence, many women who have symptoms of SUI or not seek treatment remain without resolution of symptoms.Then there is the possibility of using non-invasive radiofrequency and non-ablation in external urethral meatus in order to stimulate collagen production, as one of the pathophysiological mechanisms of stress urinary incontinence is the collagen deficit in the urethral wall. It is a randomized clinical trial and the group experimental will utilize radiofrequency and kinesiotheraphy ( clinical and in home) and the group control utilize turn off- radiofrequency and kinesiotherapy (clinical and in home). The protocol f the kinesiotherapy is the same both the group, and the protocol radiofrequency the group experimental will 5 sessions (one per week) with temperature 38ºC during 2 minutes. The group control will 5 sessions (one per week) but the radiofrequency will off but glycerin is heated, for masking for the patient, during 2 min. The result of the treatment is assessed by pad test 1 hour and have others outcomes ( quality of life- Sf-26 ans King Health- and sexual function- FSFI questionaire)

ELIGIBILITY:
Inclusion Criteria:

* 21 Women with age between 18-59 years old,
* women with diagnosis of urinary incontinence and have a Pelvic floor muscle contractility was assessed by digital palpation using the validated Modified Oxford Scale (MOS) greater than or equal to three

Exclusion Criteria:

* Patients with cognitive deficits or psychiatric illness;
* suffering from chronic degenerative neurological diseases; which have greater than 50 ml post-voiding residue ;
* sensory deficit in the genital region;
* people with pacemakers and implantable cardioverter-defibrillator and pregnant women will be excluded from the study

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-09; Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Urinary loss modification | one week, one month, two month , three month and six month
  The pad test will be held at the beginning of treatment and one week, one month, two month, three month and six month after the last session of radio frequency. The pad test it quantifies in grams urinary loss through the absorbent weighing.

SECONDARY OUTCOMES:
specific Quality of life | one week
  The quality of life will be assessed by one for specific urinary symptoms - Health King , measure with unit of the scale
Sexual Function | one week
  Will be evaluated before and after radio frequency sexual function of women, through questionary FSFI in which there is a switching station which evaluates the presence of sexual dysfunction, and there is specific scores for the domains of pain, desire, lubrication, arousal, orgasm, and satisfaction.
overall quality of life | one week
  Will be evaluated before and after radio frequency the overall quality of life - SF-36 - questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lordelo, PhD, Principal Investigator — Centro de Atenção ao Assoalho Pélvico - BAHIANA
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil